CLINICAL TRIAL: NCT05217342
Title: Peripheral Venous Pressure-Guided Decongestive Therapy in Heart Failure
Brief Title: PVP-Guided Decongestive Therapy in HF
Acronym: PERIPHERAL-HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Collaborators: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other); Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-2022-001
Record Dates: First submitted 2022-01-01; First posted 2022-02-01 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Edema; Volume Overload; Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Intervention Model Description: Two arms with a standard care control group and a peripheral pressure guided intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVP-Guided (Experimental): Peripheral venous pressure guided therapy arm
  Interventions: Drug: Diuretic therapy
- Control (Active Comparator): Standard medical therapy arm
  Interventions: Drug: Diuretic therapy

INTERVENTIONS:
Drug: Diuretic therapy — Standard diuretic therapy according to the current guidelines

SUMMARY:
The investigators hypothesize that a simple assessment of peripheral venous pressure (PVP) will better predict the diuretic need and long-term outcomes (all cause mortality, all cause rehospitalization, emergency department visits) compared to standard evaluation.

DETAILED DESCRIPTION:
I. BACKGROUND AND SIGNIFICANCE

Precise assessment of volume status is essential in diagnosis and management of diuretic therapy in patients hospitalized for heart failure (HF). Unfortunately, no clear guidelines are present for in-hospital management of congestion. Consequently, nearly half of the patients hospitalized for congestive HF are discharged with persistent congestion. This contributes to high rates of readmission and mortality.

Recently, it has been shown that a simple assessment of peripheral venous pressure (PVP) demonstrates a high correlation with central venous pressure (CVP), indicating that PVP may be useful in the standard bedside clinical assessment of volume status in HF patients to help guiding decongestive therapy.

II. THE HYPOTHESIS

The investigators hypothesize that a simple assessment of peripheral venous pressure (PVP) will better predict the diuretic need and long-term outcomes (all cause mortality, all cause rehospitalization, emergency department visits) compared to standard evaluation.

III. METHODS

1. Application for Institutional Review Board (IRB)/Ethics board approval The study will be conducted at Marmara University, Pendik Training and Research Hospital, Cerrahpaşa University Hospital, Darıca Farabi Training and Research Hospital, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, and Başaksehir Çam & Sakura Hospital, all of which are tertiary referral centers for heart failure. An IRB/Ethics board approval will be obtained from the local ethics boards.
2. Study population Patients >18 years old who were admitted with a de novo or decompensated chronic HF will be enrolled. Patients will be included regardless of ejection fraction or etiology of HF, but these will be noted as baseline variables. All patients or legal surrogate decision makers will be requested to provide a written informed consent prior to enrollment. Patients who does not consent, those with upper extremity venous pathology, those with a baseline creatinine level equal to or above 3.5 mg/dL, those with severe stenotic valvular disease and hypertrophic cardiomyopathy will be excluded.
3. Centers and Personnel The study will be undertaken at Marmara University, Pendik Training and Research Hospital, Cerrahpaşa University Hospital, Darıca Farabi Training and Research Hospital, Başaksehir Çam & Sakura Hospital and Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital.
4. Data Collection The study will start at Marmara University, Pendik Training and Research Hospital, Başaksehir Çam & Sakura Hospital, Cerrahpaşa University Hospital, Darıca Farabi Training and Research Hospital and Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, at January 1, 2022 (after the approvals from the local ethical committees are obtained).

Baseline variables Baseline variables will be collected via chart review and entered to the study form (see below).

Procedures A peripheral intravenous (IV) access, using an 18 to 22-gauge IV line, will be placed preferably to an upper extremity vein before enrollment. This line will be used to draw blood samples first. After blood samples were collected the subjects will be randomized to standard or PVP guided therapy groups. Randomization will be done using a computer-generated random allocation list. The details of demographic characteristics, symptoms, physical examination findings and drug list will be noted to a standard study form (see below).

A routine electrocardiogram and echocardiogram (including stroke volume calculated form left ventricular outflow tract size and velocity-time integral; diastolic mitral flow Doppler and mitral annular tissue Doppler measurements, inferior vena cava diameter and respiratory variation) and an 8-point lung ultrasound for total B-line count will be performed at the earliest convenience and before discharge.

After the blood samples were collected, line will be flushed carefully. PVP will be obtained by transducing a peripheral intravenous line after zeroing at the phlebostatic axis. The phlebostatic axis will be accepted as the midpoint between the anterior and posterior surfaces of the chest at the level of the fourth intercostal space meets with sternum, which is assumed to be correlated with the mid-level of the right atrium. The patient's arm will be placed parallel to the patient such that the position of the peripheral IV to be at the phlebostatic axis. Continuity of the peripheral IV line with the central venous system will be confirmed by demonstrating augmentation of the venous pressure waveform using manual or tourniquet circumferential occlusion of the extremity proximal to the catheter. If the pressure waveform failed to augment appropriately, data will not be collected, and the patient will be documented for study purposes as a technique failure. Daily fluid intake and output, weight, and biochemistry measurements, as required, will be done.

The patients in whom the first and the predischarge PVP cannot be measured due to technical issues (unable to provide upper extremity IV access, unable to confirm augmentation test) will be excluded from the study. Also, the patients requiring in-hospital intubation, high-dose inotrope or vasopressor infusion (≥10 mcg.kg-1.min-1 dopamine, dobutamine or equivalent), intraaortic balloon support, dialysis or venovenous ultrafiltration will be excluded from the study (but these patients will be included in the in-hospital analyses).

In hospital diuretic treatment will be guided by European Society of Cardiology guidelines (see below for algorithm). In standard therapy arm, the treatment and the decision of discharge will be left to physicians' discretion. In the PVP-guided arm, a PVP ≤9 mmHg will be targeted before discharge.

Outcomes The primary outcome of the study is the composite endpoint of all-cause mortality, all-cause hospitalization and all-cause emergency department visits. The secondary outcomes will include cardiovascular mortality, HF-related hospitalization, HF-related emergency department visits. These information on these outcomes will be obtained from national electronic database. The follow-up duration is planned to be limited to one-year.

Summary of patient enrollment criteria

Inclusion criteria

* Hospitalization for heart failure (de novo or decompensated chronic heart failure)
* Age >18

Exclusion criteria

* A prior history of upper extremity venous disease
* Serum creatinine ≥ 3.5 mg/dL
* Severe stenotic valvular disease
* Hypertrophic obstructive cardiomyopathy

Exclusion from long term follow-up after randomization

* Unable to obtain first and pre-discharge PVP due to technical issues (unable to access an upper extremity vein, negative augmentation test)
* In-hospital intubation
* Need for high-dose vasopressor or inotrope medications (≥10 mcg.kg.-1.min-1 dopamine, dobutamine or equivalent)
* Need for intra-aortic balloon pump support
* In-hospital need for dialysis or veno-venous ultrafiltration

Predefined secondary analyses

There will be substudies from the same cohort utilizing other analyses, as defined below:

* The correlation between predischarge PVP and long-term outcomes. A multivariable analysis will also be executed for predicting the primary end point.
* The correlation between the change in PVP during hospital stay and long-term outcomes. A multivariable analysis will also be executed for predicting the primary end point.
* The correlation between the change in PVP during hospital stay and worsening renal function, need for dialysis or veno-venous ultrafiltration.
* The comparison of the two arms in terms of worsening renal function, need for dialysis or veno-venous ultrafiltration.
* The comparison of the two arms in terms of EVEREST congestion score.
* The comparison of the two arms in terms of the days in hospital.
* The comparison of the two arms in terms of the number of repeat hospitalization.
* The relationship between venous compliance and short and long-term outcomes.

Estimated number of subjects to be submitted:

It is estimated that the enrollment of 586 participants would provide the study with a statistical power of 95% to detect a relative excess rate of 10% in primary outcome (peripheral pressure guided group 20% versus standard approach 30%) with the use of a two-sided test at the 0.05 level. Accordingly, it is expected to enroll at least 600 patients in a one-year enrollment period.

Statistical Analysis Baseline characteristics will be summarized using standard descriptive statistics. Comparisons of relevant parameters between groups will be performed by chi-square, Fisher's exact test, Mann-Whitney U, Kruskal-Wallis H test, one-way ANOVA and student t-test, as appropriate. Patients with missing values will be excluded pairwise from analyses. Kaplan-Meier analysis will be performed to determine the cumulative long-term mortality and composite outcome rates in subgroups. The mortality across groups will be compared using log-rank test. A Cox-regression model will be used to perform a survival analysis according to pre-discharge peripheral venous pressure and composite outcome. Baseline characteristics with a P value of 0.05 or less in the univariate analysis will be included and a step-down procedure will be applied for selection of final covariates. Statistical analyses will be performed with Statistical Package for Social Sciences (SPSS, version 24.0; SPSS Inc., Chicago, IL) and MedCalc Software (version 18.2.1 [Evaluation version]; MedCalc Software, Ostend, Belgium).

ELIGIBILITY:
Inclusion criteria

* Hospitalization for heart failure (de novo or decompensated chronic heart failure)
* Age >18

Exclusion criteria

* A prior history of upper extremity venous disease
* Serum creatinine ≥ 3.5 mg/dL
* Severe stenotic valvular disease
* Hypertrophic obstructive cardiomyopathy

Exclusion from long term follow-up after randomization

* Unable to obtain first and pre-discharge PVP due to technical issues (unable to access an upper extremity vein, negative augmentation test)
* In-hospital intubation
* Need for high-dose vasopressor or inotrope medications (≥10 mcg.kg.-1.min-1 dopamine, dobutamine or equivalent)
* Need for intra-aortic balloon pump support
* In-hospital need for dialysis or veno-venous ultrafiltration

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary combined end point | One year
  The difference in the combined rate of all-cause mortality, all-cause hospitalization and all-cause emergency department visits

SECONDARY OUTCOMES:
Secondary combined end point | One year
  The difference in the combined rate of cardiovascular mortality, HF-related hospitalization, HF-related emergency department visits.

CONTACTS AND LOCATIONS:
Overall Officials: Emre K Aslanger, Assoc. Prof., Study Director — Marmara University; Dursun Akaslan, MD, Principal Investigator — Marmara University; Özlem Yıldırımtürk, Prof., Principal Investigator — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital; Duygu İnan, MD, Principal Investigator — Basaksehir Cam & Sakura State Hospital; Yelda Saltan, MD, Principal Investigator — Basaksehir Cam & Sakura State Hospital
Locations (5):
- Turkey (Türkiye) (5):
  - Basaksehir Cam & Sakura State Hospital, Istanbul
  - Cerrahpasa University, Istanbul
  - Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Darıca Farabi Training and Research Hospital, Kocaeli

IPD SHARING:
Plan to Share IPD: Undecided